CLINICAL TRIAL: NCT00436254
Title: A Phase I Study of a DNA Plasmid Based Vaccine Encoding the HER-2/Neu Intracellular Domain in Subjects With HER-2/Neu (HER2) Overexpressing Tumors
Brief Title: Vaccine Therapy With Sargramostim (GM-CSF) in Treating Patients With Her-2 Positive Stage III-IV Breast Cancer or Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6532; NCI-2010-00869; RG1704001 (Other: Fred Hutch/University of Washington Cancer Consortium); NCT00194662 (obsolete NCT alias)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: HER2-positive Breast Cancer; Stage III Ovarian Epithelial Cancer; Stage III Ovarian Germ Cell Tumor; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Breast Neoplasms | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; Flow Cytometry; Immunologic Techniques; Immunoenzyme Techniques; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive pNGVL3-hICD vaccine admixed with GM-CSF intradermally once a month for 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: pNGVL3-hICD vaccine; Biological: sargramostim; Other: flow cytometry; Other: immunologic technique; Other: immunoenzyme technique; Genetic: protein expression analysis; Procedure: biopsy

INTERVENTIONS:
Biological: pNGVL3-hICD vaccine — Plasmid-based DNA vaccine, given intradermally
Biological: sargramostim — Given intradermally
  Other Names: GM-CSF; granulocyte macrophage colony-stimulating factor; Leukine; Prokine; rhu GM-CFS
Other: flow cytometry — Correlative studies
Other: immunologic technique — Correlative studies
  Other Names: immunological laboratory methods; laboratory methods, immunological
Other: immunoenzyme technique — Undergo ELIspot (correlative studies)
  Other Names: immunoenzyme techniques
Genetic: protein expression analysis — Undergo ELISA (correlative studies)
Procedure: biopsy — Undergo punch biopsy (correlative studies)
  Other Names: biopsies

SUMMARY:
RATIONALE: Vaccines may help the body build an effective immune response to kill tumor cells. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving vaccine therapy together with sargramostim may be an effective treatment for breast cancer and ovarian cancer. PURPOSE: This phase I trial is studying the side effects and identifying the best dose of vaccine therapy when given together with sargramostim in treating patients with stage III-IV breast cancer or ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the safety of intradermal administration of 3 doses of a plasmid-based DNA vaccine encoding the ICD of HER2 administered with a fixed dose of GM-CSF. II. To determine whether a plasmid DNA vaccine encoding the ICD of HER2 can elicit HER2 specific immune responses. SECONDARY OBJECTIVES: I. To determine if the dose of the plasmid-based DNA vaccine effects immunologic responses. II. To determine the persistence of DNA at the site of vaccination. OUTLINE: This is a dose-escalation study of a plasmid-based DNA (pNGVL3-hICD) vaccine. Patients receive pNGVL3-hICD vaccine admixed with GM-CSF intradermally once a month for 3 months in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up periodically for up to 15 years with primary physicians.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer: stage III or stage IV breast cancer with metastasis in remission and defined as NED (no evidence of disease); stable or healing bone disease by radiologic evaluation which may include, but is not limited to, bone scan, MRI, or PET scan documented within 90 days of enrollment to study and NED status for extraskeletal metastasis
* Ovarian cancer: stage III or stage IV ovarian cancer in first complete remission with a normal AND stable CA-125; thus, two sequential normal CA-125 values will need to be documented; a minimum of 30 days between 2 sequential CA-125 values; the most recent will be within 2 weeks of enrollment into study
* HER2 overexpression by immunohistochemistry (IHC) of 2+ or 3+ in their primary tumor or metastasis, and if overexpression is 2+ by IHC or in the absence of IHC, then patients must have documentation of HER2 gene amplification by FISH
* Eligible subjects must have completed appropriate treatment for their primary disease and be off cytotoxic chemotherapy and corticosteroids for at least 1 month prior to enrollment; patients with stage III/IV breast cancer who have completed chemotherapy and are continued on trastuzumab monotherapy are eligible; hormonal and bisphosphanate therapies are allowed
* Subjects must have a Performance Status Score (Zubrod/ECOG Scale) = 0
* All subjects must no longer be able to bear children
* Hematocrit >= 30
* Platelet count >= 100,000
* WBC >= 3,000/ul
* Creatinine =< 2.0 or creatinine clearance >= 60 ml/minute
* Serum bilirubin < 1.5 mg/dl
* SGOT < 2 x ULN
* Subjects must have recovered from major infections and/or surgical procedures and, in the opinion of the investigator, not have a significant active concurrent medical illness precluding protocol treatment or survival
* Normal ANA, anti-dsDNA and C3
* Patients on trastuzumab monotherapy must have adequate cardiac function as demonstrated by normal ejection fraction (EF) of MUGA scan or echocardiogram

Exclusion Criteria:

* Subjects cannot be simultaneously enrolled on other treatment studies
* Any contraindication to receiving GM-CSF based vaccine products
* Prior known history of cardiac disease, specifically restrictive cardiomyopathy, unstable angina within the last 6 months prior to enrollment, New York Heart Association functional class III-IV heart or symptomatic pericardial effusion
* Prior known history of pulmonary disease other than controlled asthma
* Active autoimmune disease
* Subjects cannot have active immunodeficiency disorder, e.g., HIV

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2001-10; Primary Completion 2010-03 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Safety as measured by NCI CTCAE v 3.0 | From baseline
Immune response | From baseline

SECONDARY OUTCOMES:
Impact of dose on immunologic response | From baseline to month 15
Persistence of DNA at the injection site | At 1 and 6 months after last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Mary L. Disis, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Disis MLN, Guthrie KA, Liu Y, Coveler AL, Higgins DM, Childs JS, Dang Y, Salazar LG. Safety and Outcomes of a Plasmid DNA Vaccine Encoding the ERBB2 Intracellular Domain in Patients With Advanced-Stage ERBB2-Positive Breast Cancer: A Phase 1 Nonrandomized Clinical Trial. JAMA Oncol. 2023 Jan 1;9(1):71-78. doi: 10.1001/jamaoncol.2022.5143. PMID 36326756